CLINICAL TRIAL: NCT01353469
Title: A Multicenter, Randomized, Active-controlled, Parallel-group Study to Assess the Efficacy and Safety of Insuman Comb 25 (Insulin Human) Versus Novolin® 30R Twice Daily Over 24 Weeks in Patients With Type 2 Diabetes Mellitus Who Are Under Insulin Therapy
Brief Title: Assessment of Efficacy and Safety of Insuman Comb 25 Versus Novolin® 30R Twice Daily Over 24 Weeks in Type 2 Diabetes Patients With Insulin Therapy
Acronym: Insuman-C25-CN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12059; U1111-1120-0701 (Other: UTN)
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insuman Comb 25 (Experimental): Insuman Comb 25 will be self-injected subcutaneously twice daily 30-45 minutes before breakfast and dinner. The dose will be adjusted individually by monitoring the blood glucose values and symptoms, and following China guideline.
  Interventions: Drug: Insulin human/Insuman Comb 25 (HR1799)
- Novolin® 30R (Active Comparator): Novolin® 30R will be self-injected subcutaneously twice daily within 30 minutes before breakfast and dinner. The dose will be adjusted individually by monitoring the blood glucose values and symptoms, and following China guideline and the package insert of Novolin® 30R
  Interventions: Drug: Insulin human/Novolin® 30R

INTERVENTIONS:
Drug: Insulin human/Insuman Comb 25 (HR1799) — Pharmaceutical form:Suspension
  Route of administration: Subcutaneous
  Arms: Insuman Comb 25
Drug: Insulin human/Novolin® 30R — Pharmaceutical form:Suspension
  Route of administration: Subcutaneous
  Arms: Novolin® 30R

SUMMARY:
Primary Objective:

To compare the efficacy of Insuman Comb 25 versus Novolin® 30R on HbA1c reduction during a 24-week treatment period in patients with type 2 diabetes mellitus.

Secondary Objectives:

* To assess the effects of Insuman Comb 25 versus Novolin® 30R in patients with type 2 diabetes mellitus on fasting plasma glucose (FPG)
* To assess the safety and tolerability of Insuman Comb 25 versus Novolin® 30R in patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
The study duration per patient is about 27 weeks (up to 2 weeks screening + 24 weeks open-label treatment + 1 week follow-up).

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus patients, as defined by World Health Organization (WHO), diagnosed for at least 1 year at the time of screening visit who are under premix insulin therapy, with or without oral anti-diabetic drug (OAD)
* Signed written informed consent

Exclusion criteria:

* HbA1c <7% or HbA1c >10% at screening
* No self-monitoring of blood glucose within 3 months prior to screening visit
* Premix insulin treatment for less than 3 months. Insulins other than premix insulin treatment within 3 months prior to screening visit
* In case of treatment with OAD, treatment with a stable OAD dose and regimen for less than 3 months prior to screening visit

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to the end of treatment | 24 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose from baseline to the end of treatment | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- China (23):
  - Investigational Site Number 156024, Beijing
  - Investigational Site Number 156010, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156033, Changchun
  - Investigational Site Number 156017, Changchun
  - Investigational Site Number 156005, Changsha
  - Investigational Site Number 156021, Chengdu
  - Investigational Site Number 156006, Chongqing
  - Investigational Site Number 156032, Hangzhou
  - Investigational Site Number 156007, Harbin
  - Investigational Site Number 156020, Hefei
  - Investigational Site Number 156016, Nanjing
  - Investigational Site Number 156018, Nanjing
  - Investigational Site Number 156002, Shanghai
  - Investigational Site Number 156023, Shanghai
  - Investigational Site Number 156031, Shanghai
  - Investigational Site Number 156004, Shanghai
  - Investigational Site Number 156027, Shenyang
  - Investigational Site Number 156029, Suzhou
  - Investigational Site Number 156025, Tianjin
  - Investigational Site Number 156003, Wuhan
  - Investigational Site Number 156008, Xi'an
  - Investigational Site Number 156009, Xi'an